

# **PROTOCOL**



### Full/long title of the project:

A study to explore the feasibility and efficacy of Group Traumatic Episode Protocol (GTEP) for reducing trauma symptoms following a traumatic birthing experience.

#### Short title/acronym

The efficacy of GTEP for birth trauma.

#### Sponsor:

University of Birmingham

research governance @contacts.bham.ac.uk

#### Protocol version number and date

| Protocol version number: | 1.1 |
|--------------------------|------------|
| Protocol version date: | 14/03/2025 |

#### Research reference numbers

| IRAS number: | 341922 |
|-------------------------|-----------|
| Sponsor/RG number: | RG_24-029 |
| REC reference number: | |
| Public registry number: | |
| Funder number: | |

This protocol has regard for the HRA guidance.



### Signature page

The undersigned confirm that the following protocol has been agreed and accepted and that the CI agrees to adhere to the signed University of Birmingham's sponsorship CI declaration.

I agree to ensure that the confidential information contained in this document will not be used for any other purpose other than the evaluation or conduct of the investigation without the prior written consent of the Sponsor

I also confirm that I will make the findings publicly available through publication or other dissemination tools without any unnecessary delay and that an honest accurate and transparent account of the project will be given; and that any discrepancies from the project as planned in this protocol will be explained.

| Full project title: | A study to explore the feasibility and efficacy of Group Traumatic Episode Protocol (GTEP) for reducing trauma symptoms in individuals following a traumatic birthing experience. |
|---|---|
| Protocol version number: | v 1.1 |
| Protocol version date: | 14/03/2025 |

| Chief Investi | igator (CI) |
|---------------|---------------|
| Name: | Grace Rodgers |
| Date: | 08/07/2024 |
| Signature: | |

#### Sponsor statement

Where the University of Birmingham takes on the sponsor role for protocol development oversight, the signing of the IRAS form by the sponsor will serve as confirmation of approval of this protocol.



## Table of contents

| Title pag | e | 2 |
|---|---|---|
| Full/lo | ng title of the project | 2 |
| Short | title/acronym | 2 |
| Protoc | col version number and date | 2 |
| Resea | rch reference numbers | 2 |
| Signatur | e page | 3 |
| Spons | or statement | 3 |
| Table of | contents | 4 |
| Key cont | acts | 6 |
| Project s | ummary | 6 |
| Funding | and support in kind | 8 |
| Role of s | ponsor and funder | 8 |
| Roles & ı | responsibilities of management committees/groups & individuals | 8 |
| Patien | t & public involvement group | 8 |
| Protocol | contributors | 8 |
| Key word | ds | 8 |
| Project f | low chart | 9 |
| Protocol | | 10 |
| 1. | 13 | |
| 2. : | 13 | |
| 3. | 14 | |
| 4. | 14 | |
| 4.1. | 14 | |
| 4.2. | 16 | |
| 5. 3 | 16 | |
| 6. 2 | 20 | |
| 7. 2 | 21 | |
| 7.1. | 21 | |
| 7.1. | 1. 21 | |
| 7.1. | 2. 21 | |
| 7.2. | 22 | |
| 7.2. | 1. 22 | |
| 7.2. | 2. 22 | |
| 7.3. | 23 | |
| 7.3. | 1. 23 | |
| 7.3. | 2. 23 | |



9. 24

10. 24

10.1. 26

10.2. 26

10.2.1. 27

10.2.2. 27

10.3. 27

10.4. 27

10.5. 28

10.6. 28

10.7. 29

10.8. 29

10.9. 29

11. 29

11.1. 29

11.2. 29

12. 30

13. 34

13.1. 34

13.2. 48



# Key contacts

| Role/function | Role and Organisation | Contact details |
|---|---|---|
| Dr Rachel Strachan - Principal<br>Investigator and External Supervisor | Consultant Clinical Psychologist, Black<br>Country Healthcare NHS Foundation<br>Trust | rachel.strachan@nhs.net |
| Grace Rodgers - Chief Investigator | Doctoral student, University of Birmingham | gxr327@student.bham.ac.uk |
| Dr Alice Welham - Co-Investigator and<br>Internal Supervisor | Clinical Psychologist and Associate<br>Professor, University of Birmingham | a.welham@bham.ac.uk |
| Habibah Zeb — Co-Investigator | Assistant Psychologist, Black Country<br>Healthcare NHS Foundation Trust | habibah.zeb@nhs.net |

## Project summary

| Project Title: | A study to explore the feasibility and efficacy of Group Traumatic Episode Protocol (GTEP) for reducing trauma symptoms following a traumatic birthing experience. |
|---|---|
| Short Title: | The efficacy of GTEP for birth trauma. |
| Research question/aim: | This study aims to evaluate the feasibility and efficacy of GTEP for reducing trauma symptoms (measured by the PCL-5 and City BiTS) for individuals following a traumatic birthing experience. A secondary aim is to evaluate the efficacy of GTEP in improving parental wellbeing (measured through the CORE-10) and parent-infant bonding (measured through the PBQ) following a traumatic birthing experience |
| | This study aims to help to address a current gap in literature, contribute to the growing evidence base for GTEP and allow more individuals to access appropriate and effective support within clinical services. This may potentially reduce waiting times for psychological interventions within secondary care services (if an effective group intervention is able to be offered). |
| Project Design: | This study will use a pre-post design, with outcome measure questionnaires completed at two time points (before and after the GTEP intervention, T1 and T8). |
| | In addition, the PCL-5 outcome measure questionnaire will be given at 8 time points (i.e., during the pre-intervention home visit, before |



sessions 2, 3, 4, 5, 6 and 7 and during the postintervention follow-up). Participants will be offered 6 sessions: Session 1 – Pre-intervention appointment at participant's home. Sessions 2, 3, 4, 5, 6 and 7 – GTEP sessions completed via Zoom. Session 8 - Post-intervention follow-up (either at participant's home or via phone call). This design was chosen as we want to know the impact of the GTEP intervention in reducing trauma symptoms, as well as improving parental well-being and parent-infant bonding. The administration of pre-post outcome measures will allow us to track any significant changes in scores. A study feasibility measure (Weiner et al., 2017) will also be administered to evaluate the feasibility of the intervention for this population. Participants: Participants will be recruited via the Black Country Perinatal Mental Health Service (BCPMHS) who are self-reporting trauma symptoms related to a traumatic birthing experience within the last 18 months. All eligible participants (according to the inclusion/exclusion criteria) will be offered to take part in the group. All potentially eligible participants (identified from the BCPMHS) will be contacted via phone call to discuss the research project and GTEP group and gain verbal consent to send them the PIS and Consent Form via email/text message system (dependent on individual preference). Participants who express an interest in taking part will then be offered a 1:1 home visit (this is session 1 of the intervention). During this visit, the group/project will be discussed further and eligibility for the group will be determined. The participant will also have the opportunity to ask any questions they have, and outcome measure data will be collected. **Planned Recruitment Target:** We are hoping that the group will be run on a rolling basis, with approximately 5 participants in each group. We will continue to collect outcome measure data until the appropriate number of participants have been reached. A priori power analysis was conducted using G\*Power for a minimum sample size calculation. Results showed that to achieve 80% power for detecting a medium effect size, using a significance level of 0.05, a sample size of 28 will be adequate.



| Follow-up Duration: | Participants will be offered a post-intervention follow-up session 2-6 weeks after the final online GTEP session. This can be offered as a virtual appointment or home visit depending on the participant's preference. The final outcome measures will be completed during this session (T8). |
|---|---|
| Planned study period: | The planned study period will run between October 2024 – September 2026. |

### Funding and support in kind

This is a doctoral project as part of the Doctorate in Clinical Psychology (DClinPsy) and therefore no external funding has been secured. Any costs incurred will be covered by the University of Birmingham.

### Role of sponsor and funder

The project is being sponsored by the University of Birmingham.

The research team named above hold responsibility for the project design, conduct, data analysis and interpretation, manuscript writing and dissemination of results.

### Roles & responsibilities of management committees/groups & individuals

There are no other committees, groups or individuals involved in the project beside those named above and the sponsorship from the University of Birmingham.

#### Patient & public involvement group

Service users from the BCPMHS have been involved in a trial GTEP group to explore initial acceptability of the group. Following feedback from the service users, the structure of the group has been changed and the number of online GTEP sessions has been changed from four to six, to allow more time for stabilisation, education about the group and for group members to get to know each other.

The research team has also informally sought feedback from other services who have previously conducted GTEP groups through the GTEP Special Interest Group (SIG). This has allowed the research team to understand what has worked well previously and gather ideas for this current group.

#### Protocol contributors

The protocol contributors are:

- Dr Rachel Strachan (PI) (External to UoB)
- Dr Alice Welham (Co-Investigator)
- Grace Rodgers (CI)
- Habibah Zeb (Co-Investigator) (External to UoB)

These individuals form the research team involved in this project.

### Key words/Abbreviations

| T1, T2, T3, T4, T5, T6, T7 and T8 | Time point 1, time point 2, time point 3, time point 4, time point 5, time point 6, time point 7 and time point 8 |
|---|---|
| PCL-5 | PTSD Checklist for DSM-5 |



| City BiTS | City Birth Trauma Scale |
|-----------|--------------------------------------------------|
| CORE-10 | Clinical Outcomes in Routine<br>Evaluation 10 |
| PBQ | Postpartum Bonding Questionnaire |
| GTEP | Group Traumatic Episode Protocol |
| CI | Chief Investigator |
| PI | Principal Investigator |
| BCPMHS | Black Country Perinatal Mental<br>Health Service |



### Project flow chart

This flowchart describes the procedure for the research study. We are planning to continue the GTEP group on a rolling basis and collect outcome measure data until an appropriate number of participants have been recruited. It is anticipated that this procedure will be the same for all groups.





As the research team member completing the 1:1 review session is also a member of the clinical team cofacilitating the GTEP group within the BCPMHS, they will be able to assess whether the participant can be



discharged from the BCPMHS psychology team or be added to the waiting list for 1:1 work. They will also be able to discuss this with other members of the psychology team within the BCPMHS if needed. It is part of standard care for participants to be reviewed following a psychological intervention, and the participants usual care within the BCPMHS will not be affected if they are discharged from the psychology team. They will still be able to access support from other professionals within the team, if this is required and appropriate.

The waiting list for 1:1 work forms part of the standard care within the BCPMHS psychology team.



#### **Protocol**

#### 1. Background

It is estimated that up to 15.7% of individuals will experience some trauma symptoms following childbirth, with 4-6% developing Post-Traumatic Stress Disorder (PTSD-UK). Research has found there to be an increased risk of postpartum depression, postpartum psychosis and anxiety following a complicated or traumatic childbirth (Ertan et al., 2021), along with reduced parent-infant bonding at 1, 6 and 12-months postpartum (Kjerluff et al., 2021). Suicide has been found to be the leading cause of direct maternal death between 6-12 months postpartum (MBRRACE-UK, 2023), thus demonstrating a need for both clinical and research focus in this area. Furthermore, parents of babies admitted to a neonatal unit have been found to experience significant trauma symptoms, depression, anxiety and stress (Dickinson et al., 2022), as well as high prevalence of sleep disturbances and fatigue (Busse et al., 2013), suggesting that additional experiences surrounding the birth, not just the childbirth itself, can be traumatic.

Group Traumatic Episode Protocol (GTEP) is a version of Eye Movement Desensitization and Reprocessing (EMDR) developed by Shapiro (2013), to be used in group settings. Individual EMDR has been found to be effective at reducing PTSD symptoms at 6-weeks postpartum (Chiorino et al., 2020), but there is no research to date exploring the efficacy of GTEP for trauma symptoms related to birth. There is a growing evidence base for the efficacy of GTEP in other populations and it has been found to reduce trauma symptoms in a refugee population, adult cancer patients and healthcare professionals (Lehnung et al., 2017; Yurtsever et al., 2018; Roberts, 2018; Tsouvelas et al., 2019; Farrell et al., 2023; Pink et al., 2022). Given the prevalence of birth trauma and the subsequent detrimental consequences on parental mental health, this study hopes to add to the growing evidence base and if found to be effective, allow more individuals to access appropriate support more quickly.

#### 2. Rationale

This research will aim to evaluate the efficacy of GTEP for individuals who have experienced birth trauma. As there is no existing research investigating this, there is a need for this study to address



this gap in the literature. Given the prevalence of traumatic birthing experiences, the subsequent effects on parental wellbeing, and the demand on specialist perinatal services, this research will also help inform the development of these services and allow more individuals to access appropriate support more quickly. This is especially important in this population given the detrimental effects of birth trauma on postnatal mental health in women/birthing people. Furthermore, research has found that poor parental mental health can affect a child's attachment, and their cognitive, social and emotional development (Manning and Gregoire, 2009), with maternal anxiety being associated with poor educational attainment (Ayano et al., 2022).

Although individual EMDR has been found to be effective for reducing birth trauma symptoms and there is a strong evidence base, this research will be the first to explore GTEP (a form of group EMDR) with this population and will likely have important clinical implications in informing the way that trauma symptoms related to a traumatic birthing experience are treated within mental health services.

#### 3. Theoretical framework

This piece of research sits within the growing evidence base for the use of GTEP in clinical settings. GTEP is a group version of the Recent Traumatic Episode Protocol (R-TEP) developed by Shapiro and Laub (2008), which conceptualises that recent traumatic events have not had time to conceptualise and remain fragmented for an individual. GTEP aims to keep many of the R-TEP principles (e.g., history taking, preparation and stabilisation, and episode processing). It has been found to be effective with refugee populations, adult cancer patients, healthcare workers, female victims of intimate partner violence and genocide survivors, but no research to date has explored its efficacy within a perinatal population. Therefore, this research will aim to address this gap in literature.

#### 4. Research question/aims

This research aims to evaluate the feasibility and efficacy of GTEP for reducing trauma symptoms in individuals who have had a traumatic birthing experience. In addition, it will also explore the effectiveness of GTEP in improving parental wellbeing and the parent-infant relationship.

#### 4.1. Objectives

| Objectives | Outcome Measures (to achieve this |
|------------|-----------------------------------|
| | objective) |



| Primary Object | :tive: |
|----------------|--------|

To assess any changes in trauma symptoms following participation in the GTEP intervention for individuals who have had a traumatic birthing experience.

Trauma symptoms will be measured using the PTSD Checklist for DMS-5 (PCL-5) (Blevins et al., 2015).

Childbirth-specific trauma symptoms will be measured using the City Birth Trauma Scale (City BiTS) (Ayers et al., 2018).

These measures have been validated for use.

The PCL-5 will be completed at 8 time-points:

- During pre-intervention home visit (session 1 of the intervention) (T1)
- Before session 2 of the intervention (T2)
- Before session 3 of the intervention (T3)
- Before session 4 of the intervention (T4)
- Before session 5 of the intervention (T5)
- Before session 6 of the intervention (T6)
- Before session 7 of the intervention (T7)
- During the post-intervention followup session (T8)

The City BiTS scale will be completed at T1 and T8.

#### **Secondary Objective:**

To assess any changes in the wellbeing of the birthing parent following the GTEP intervention. Wellbeing will be measured using the Clinical Outcomes in Routine Evaluation 10 (CORE-10) (Barkham et al., 2013).

The CORE-10 will be completed at T1 and T8.

#### **Secondary Objective:**

To assess any change in parent-infant bonding following the GTEP intervention.

Parent-infant bonding will be measuring using the Parental Bonding Questionnaire (PBQ) (Brockington et al., 2001)

The PBQ will be completed at T1 and T8.

#### **Secondary Objective:**

To assess the feasibility of the GTEP intervention for a birth trauma population.

Feasibility will be measured through using the Acceptability of Intervention Measure (AIM), Feasibility of Intervention Measure (FIM) and Intervention Appropriateness Measure (IAM) (Weiner et al., 2017). These



| BIRMINGHAM | |
|---|---|
| | questions will be asked at the beginning of each session from T2 – T8. |
| | These questions will also be asked to facilitators, before and after the intervention. |
| | Open-ended qualitative questions will also be asked during the post-intervention follow-up session. |

#### 4.2. **Outcome**

Potential outcomes of this study include:

- To contribute to the growing evidence base for the use of GTEP in clinical settings, with individuals who have experienced a traumatic event.
- Be the first study to explore the efficacy of GTEP for individuals with a traumatic birthing experience, within a secondary care service.
- Help to inform the treatment for individuals who have had a traumatic birthing experience.
- Enable more individuals to access treatment in a timely way as group interventions can be offered more quickly than individual interventions. This, in turn, could also reduce pressure on specialist services as the interventions could be offered within maternity and primary care (e.g., Talking Therapies). This could result in less referrals being made into secondary care services and a reduction in waiting times within these services.

### 5. Design and methods of data collection and data analysis

<u>Project Design:</u> This study will adopt a pre-post experimental design to explore the efficacy of GTEP on reducing trauma symptoms for individuals who have experienced a traumatic birthing experience. The outcome measures will be completed before and after the intervention, to determine any changes.

Participants will be recruited from the BCPMHS, which is part of the Black Country Healthcare NHS Foundation Trust. Potentially eligible participants (i.e., those reporting trauma symptoms following a birthing experience in the last 18 months), will be identified at any point during their care with the BCPMHS. For example, during their initial assessment with the service, during a psychology drop-in session with members of the MDT, during an appointment with another discipline within the team. These individuals will be asked by the clinician conducting the assessment / appointment / lead clinician involved in their care whether they are willing to be contacted by a member of the research team to discuss the research study.

Individuals will then be contacted by a member of the research team via telephone to discuss the research project/GTEP group. During this discussion, information will be provided about the group and research study and the research team member will check eligibility regarding access to technology and internet access. Verbal consent to send the PIS and consent form via Accurax will be sought and this verbal consent will be documented in their clinical notes. A member of the clinical team will have already reviewed the individual's clinical notes to determine initial eligibility (e.g., age, symptoms of birth trauma



following a birth within the last 18 months, English language speaking). If the individual does not have access to technology but would like to engage in the group, then we can put them in contact with the Digital Inclusion Project within the Black Country Healthcare NHS Foundation Trust to help with this. Following this telephone call and if the individual expresses an interest in the study, they will be sent a link via Accurax to an MS Forms containing the Participant Information Sheet (PIS) and Consent Form. Accurax has been approved for use by the BCPMHS. A home visit will then be arranged with the participant and consent will be taken at the beginning of this appointment to ensure they have consented. If they do not consent, then the session will end and no research activities will occur. The PIS and consent form will have been sent via Accurax prior to this session for the participant to read and process, but paper forms can also be taken to the session if necessary.

During this session (providing that consent has been obtained at the beginning of the appointment), the staff member will determine whether the individual is able to engage in a group therapy based on their clinical presentation. For example, individuals presenting with high levels of dissociation and/or anxiety may not be suitable for the group. This staff member will be a member of the psychology clinical team (likely to be the Trainee Clinical Psychologist on placement with the BCPMHS) so will be appropriately qualified to determine eligibility. They will also be able to discuss with other members of the psychology team should there be any questions or concerns about participant suitability. Eligibility according to any inclusion/exclusion criteria that have not yet been covered will also be established. The consent form will be uploaded to Rio once completed, so therefore will remain as part of their record. However, should the participant not be deemed suitable for the group at a later date (e.g., during this visit), then a progress note will be added to Rio explaining this and the reason for it. As questionnaire data will have been completed on Rio, this will also remain on their record.

The outcome measures for T1 will be completed during this home visit, on a laptop with the team member. These outcome measures will be completed and stored on the individual's clinical record (using the system Rio). There can be a second staff member not involved in the group to help support the completion of these measures, if necessary.

It is anticipated that the group will then be completed on a rolling basis until an appropriate number of participants and data have been gathered.

Participants will be offered six online group GTEP sessions conducted via Zoom (sessions 2 – 7 of the intervention). Either a UoB or BCPMHS Zoom account will be used for this. No personal accounts will be used and the sessions will not be recorded. These sessions will be conducted by 2-3 Clinical Psychologists (depending on numbers in the group) within the BCPMHS who have been trained in EMDR and GTEP. There will also be a Trainee Clinical Psychologist present within the group, who will be an 'emotional support person' and provide additional support in break out rooms/phone call after the session should a participant require this. All participants will be offered a catch-up phone call between sessions, regardless of whether they have reported distress during the session. Each session will be



1.5 hours long. The initial sessions will be focused on the group participants getting to know each other, psychoeducation about trauma, preparation for processing work, basic grounding and stabilisation techniques. This will likely involve breathing techniques and imagery techniques, such as 'safe place' imagery. The following sessions will focus on the processing of the traumatic memory, using GTEP principles. This processing will focus on different 'Points of Disturbance' (PODs) associated with the traumatic memory. The exact processing will be unique to each individual and dependent on their own PODs. This session structure will depend on clinical judgment and group presentation and will respond to the needs of the group as required regarding the content of the sessions. For example, if it is felt that more than two sessions are needed for grounding and psychoeducation, then there will be flexibility within the session plans to do this.

For any processing sessions, the script from the GTEP protocol will be followed (see Appendix 1).

The participants will then be offered a 1:1 follow-up review between 2-6 weeks after session 7 (the final GTEP session). This will form session 8 of the intervention and will include a debrief about the intervention, complete the outcome measures for T8 and determine if any further support is needed.

Feasibility questions about the participant's experience of being part of the group will also be asked, and written responses recorded, during this session. We will use Weiner et al's (2017) Acceptability of Intervention Measure (AIM), Intervention Appropriate Measure (IAM) and Feasibility of Intervention Measure (FIM) to do this. Responses are provided on a Likert scale where I = Completely Disagree and 5 = Completely Agree. The questions are as follows:

#### AIM:

- I. "I like the intervention."
- 2. "I welcome the intervention."
- 3. "This intervention is appealing to me."
- 4. "I approve of this intervention."

#### FIM:

- 1. "This intervention seems possible to implement."
- 2. "The intervention seems doable for me."
- 3. "The intervention is easy to use."
- 4. "I can see myself continuing to use this intervention."

#### IAM:

- I. "This intervention seems like a good fit for me."
- 2. "This intervention seems suitable for my needs."
- 3. "This intervention seems appropriate for my situation."
- 4. "This intervention makes sense to me."



We will also ask two open-ended qualitative questions, which are: "What worked well about the GTEP intervention" and "Is there anything you would have changed about the GTEP intervention?". The Likert scaled questions will be asked at the beginning of each session (from session 2 onwards). This will mean we can capture the data of participants, should they drop-out partway through the intervention. The open-ended qualitative questions will only be asked during session 8, the post-intervention follow-up.

These will be written responses, and no audio recording will be conducted. Asking participants questions about their experience of psychological interventions should form part of best-practice care, and so this process will not deviate from feedback that would be gathered as part of care as usual. This information may be used in later qualitative analysis related to feasibility.

Should a participant not complete the group, or if they are considering discontinuing, they will be given the opportunity to give feedback related to this. Again, this will be written, and no audio recording will be conducted. This information may be used in later qualitative analysis related to feasibility.

Group facilitators will also be asked to report on their experiences of running the group. The same questions as above (the AIM, FIM and IAM) will be asked to facilitators. These will be asked before and after administering the intervention.

As per the authorship, there may be minor changes made to the questions to make them appropriate for the group being asked (i.e., participants or facilitators).

Facilitators will also be asked open-ended qualitative questions on their experience of the group, which will include the questions of "What worked well in running the GTEP intervention?" and "Is there anything you would change about the intervention?" Again, this information may be used in later qualitative analysis related to feasibility.

The written responses will not contain any identifiable information. Responses will be matched to participant ID numbers. The information will be stored on a secure shared drive within the BCPMHS and then be securely transferred to the UoB Research Data Store for analysis, if required.

In regard to usual care, the study will offer an additional intervention (GTEP) to the usual care for women under the BCPMHS. Standard care would involve these women being added to a waiting list to receive 1:1 psychological support for birth trauma. Instead, if appropriate and eligible, they will be offered the group instead. As explained previously, if the participant declines to attend the group or they do not meet inclusion/exclusion criteria, they will be offered the standard care of 1:1 work and added to the waiting list for this. Similarly, if the participant drop-outs of the group partway through or it is determined that they require further support once the group has finished, then they will be offered the usual care of 1:1 work, and the added to the waiting list for this.

#### Data Collection:

All outcome measures (PCL-5, CBTS, CORE 10 and PBQ) will be completed during session one of the intervention - the 1:1 home visit (T1), by one of the group facilitators. These will be completed on either Rio (the clinical records system used by the BCPMHS) or an MS



Forms, using the team member's laptop. The PCL-5 will be repeated before sessions 2-7 of the GTEP group (T2 - T7). These will be completed electronically using MS Forms and participants will be sent a link to this. The PCL-5 will be completed again during the post-intervention home visit (T8), using either Rio or MS forms.

All other outcome measures will be repeated only at the post-intervention follow-up session (T8), either via Rio or using MS Forms.

The outcome measure data will not contain any identifiable information, and be linked only by participant ID.

Data will be analysed at the University of Birmingham. Research team members external to UoB will not be involved in data analysis. Data analysis will be completed by Grace Rodgers, Trainee Clinical Psychologist and Dr Alice Welham, Clinical Psychologist/Associate Professor, both internal at UoB.

#### Data analysis:

Data analysis will be completed using Statistical Package for Social Sciences (SPSS) software. Quantitative data analysis will include a pre-and-post-intervention comparison scores at both an individual and a group level. Reliable Change Index (RCI) analysis will be employed to examine differences on an individual level. Pre-to-post change on a group level will be examined using either a bootstrapped paired samples t-test or a matched pairs Wilcoxon (depending on N and properties of data distribution). There will likely be an emphasis on effect sizes over statistical significance, especially given the possible small sample size. Further analyses will be conducted where possible/appropriate to explore whether demographic factors (e.g., age, ethnicity) or initial outcome measure scores (e.g., the 'severity' of symptoms) influenced or predicted any observed changes in scores (e.g., correlational or between-subgroups analyses of change scores).

Depending on the results, the group may be split into "responders" and "non-responders" based on the RCI analysis.

This will potentially then allow appraisal of the degree to which factors like age, initial questionnaire scores or time since trauma are statistically related to whether the group is associated with a reliable effect. This may involve, for example, Mann-Whitney or between-participant t tests (e.g., comparing responders and non-responders on age or initial PCL-5 score). We acknowledge the increased possibility of Type 1 errors due to multiple tests. Whilst we intend to emphasise effect sizes over statistical significance, we will consider this within our analysis. Bonferroni correction may be too conservative within this project, we will report significance of any effects at multiple levels of alpha and consider them within the context of the analyses performed.

Descriptive statistics will also be used where appropriate.

Qualitative analysis may be conducted related to the feasibility questions outlined above.

#### 6. Project setting

This study will be conducted within the BCPMHS. This setting enables access to individuals who have experienced a traumatic birthing experience and require a psychological intervention to address this. Participants will be recruited at any point during their care with the BCPMHS. Session 1 of the intervention will take place in the participant's homes and the



GTEP group (session 2-7) will be conducted via Zoom. The post-intervention follow-up (session 8) will either be conducted on the telephone or at the participant's home, depending on their preference.

All participants will continue to access treatment-as-usual from other disciplines within the perinatal service (e.g., psychiatry, nursery nurse).

#### 7. Participant recruitment

This project will recruit individuals who have had a traumatic birthing experience (the birth itself, the postnatal hospital stay, and/or any neonatal admissions) within the last 18 months. They will be identified through self-reported trauma symptoms (e.g., flashbacks, nightmares) at initial assessment within the service (usually with a mental health clinician), or at a subsequent appointment with any staff member within the service.

#### 7.1. Eligibility criteria:

#### 7.1.1. Inclusion criteria

- Aged between 18-65 years.
- Currently under the Black Country Perinatal Mental Health Service
- Experiencing self-reported trauma symptoms related to a birthing experience within the last 18 months (this includes the birth itself, the postnatal hospital stay, and/or any neonatal admissions).<sup>1</sup>
- Access to technology (e.g., laptop, internet connection) to be able to access the online group.<sup>2</sup>
- Access to a confidential space within their home, and childcare for their baby/any other existing children.
- Proficient levels of English Language to engage with the group.
- Ability to engage in group therapy based on clinical presentation.
- Capacity to consent to engage in the GTEP group and research study.

#### 7.1.2. Exclusion criteria

- Pregnant people.
- Women/birthing people whose baby is no longer under their care.
- Severe and enduring mental health presentations (i.e., diagnosis of bipolar, psychosis and/or schizophrenia.<sup>3</sup>

¹It was decided to include individuals experiencing trauma symptoms related to the postnatal hospital stay/neonatal admission as well as the birth itself, as clinical experience has shown that individuals often report these aspects of the birthing experience to be the most traumatic. This will allow more individuals to be recruited into the study.

<sup>&</sup>lt;sup>2</sup> Where this is not available, we are able to refer to a digital inclusion project within the Black Country NHS Foundation Trust who will be able to provide support.

<sup>&</sup>lt;sup>3</sup> This has been implemented due to the risk of a trauma intervention causing a deterioration in the participants' mental health and the possible difficulties of managing risk within a group setting. While there is no current evidence base for this intervention, it feels safer to continue supporting these individuals on a 1:1 basis.



Significant sensory impairment (e.g., needing a British Sign Language interpreter).

In regard to the group facilitators, these will be psychological professionals (likely Clinical Psychologists) working with the BCPMHS who have received training on EMDR and GTEP. They will be approached by a member of the research team to discuss being involved in research study. An initial conversation about the study will then be arranged, either in-person or over a phone call / online video conferencing platform. They will also be given the facilitators PIS to read at this point (either in person or sent via MS Forms). Following this conversation, if they are happy to be involved, a consent form will need to be signed and returned within two weeks of the initial conversation.

Given the nature of the GTEP and that fact it is forming part of clinical practice / therapeutic offering within the psychology team in the BCPMHS, should facilitators not want to be involved in the research study element of the group (i.e., answering questions regarding the group's feasibility), they will likely still be able to be a part of facilitating the group clinically.

The hard copies or MS Forms of the consent forms will also be kept as part of the research file / data, which will be kept at the University of Birmingham for 10 years.

#### 7.2. Sampling

#### 7.2.1. Size of sample

We are hoping to recruit approximately five participants per group. A priori power analysis was conducted using G\*Power for a minimum sample size calculation. Results showed that to achieve 80% power for detecting a medium effect size, using a significance level of 0.05, a sample size of 28 will be adequate. The groups and data collection will aim to be continued on a rolling basis until a suitable number of participants have been recruited and data has been collected. The planned sample size is 28 based on the above power calculation.

#### 7.2.2. Sampling technique

All eligible participants (according to the above criteria) will be offered to take part. Participants can be identified at any point during their time with the BCPMHS. Some participants may be identified during their initial assessment into the service. The assessing clinician, from the BCPMHS (the direct care team), will identify any potential participants (i.e., reporting a traumatic birthing experience within the last 18 months) during this assessment. Anyone that appears initially eligible will be asked during this initial assessment if they would be happy for a member of the research / clinical team to call them to discuss the group/research project. Verbal consent will be gained from the individual for this contact, and consent to use their contact details for this purpose. All assessments are discussed within the MDT meeting and if deemed potentially appropriate for the group / research study, a team member will contact them via phone to discuss the research study and send a link to the PIS and consent form.

Contact numbers will be accessed via the clinical records system, by a member of the clinical team. As the research team will also be working within the BCPMHS they will be able to access participant's contact details, as the individual will have consented for the team to have their contact details on referral to the service. It will also be documented on the initial



assessment clinical note that a discussion was had with the individual about the potential for the GTEP group / research project involvement.

Additionally, participants may also be identified during other points in their care. For example, they may be identified during a psychology consultation drop-in session, during an MDT discussion that happens within a team meeting, following an appointment with another discipline with the team. If a potential participant is identified in this way, the staff member from the BCPMHS who has had previous contact with the individual (e.g., psychiatry, nursery nurse, care co-ordinator), will have a discussion with the individual about the GTEP group. As per best practice, they will be asked if they are happy for a member of the team involved in the project to contact them to discuss this further. If happy, the above process will be followed by contacting via phone and sending a consent form and PIS.

#### 7.3. Recruitment

Participants will be recruited via the Black Country Perinatal Mental Health Service. Eligible participants will be identified either from an assessment / by other team members within the service, at any point during the care under the BCPMHS (as described above). If they are interested in the study/happy for a research team member to contact them via phone, then they will receive a phone call to discuss the project in more detail. If they are still interested, a link to a PIS/consent form will be sent following this phone call, and the consent form will be completed at the beginning of the home visit to ensure the participant has given appropriate consent for this session to take place.

#### 7.3.1. Sample identification

Participants will only be identified and recruited from the BCPMHS. Staff members within the perinatal service will identify potential participants during an initial assessment and further information (including consent form and PIS) will be provided in a phone call with a member of the clinical/research team. Eligible participants might also be identified from the psychology waiting list or by other clinicians / during other appointments within the BCPMHS, as described above.

Participants will not be provided with any financial incentive for participation in the study.

#### 7.3.2. Consent

Informed consent will be obtained prior to the participant completing any activities that are for the purpose of the research study. Information about the study will be provided via phone call following identification of them being a potentially eligible participant (if they have confirmed their interest in the group/study). Following this phone call, participants will be sent a link to an MS Forms with the PIS and Consent Form (if they are still interested) for them to read and process the information. A home visit will be arranged, and consent will be taken in-person at the beginning of the session (before any further activities take place) to ensure the participant has given appropriate consent. If they do not consent, the session will be ended, and no further activity will take place.

Participants have a right to withdraw at any time during the research study. If they choose to withdraw, they will be added onto the waiting list for a psychology assessment and/or therapeutic intervention, as appropriate (depending on where they were in the service



referral process at time of recruitment). This is the procedure of standard care within the service.

All participants will continue to receive 'treatment as usual' within the perinatal service whether they engage with the research study or not (e.g., access to other members of the multidisciplinary team, psychiatry, nursery nurse etc).

If a participant withdraws, as they would have consented to the procedures they had already undergone, data will be retained and used in analysis if appropriate.

#### **Translation for participants**

Participants will be required to have a proficient level of verbal English to be able to access and engage with the group. We will not be able to provide a translator during the group, so part of the pre-assessment visit will involve determining that the participant has proficient levels of English in order to engage with the group. This will be done through checking their understanding of the verbal information being provided and assessing how far they are able to engage in conversations in English.

Participants will not be excluded for not having written English ability (e.g., being unable to read/write). In this instance, information would be delivered verbally/in pictures rather than written. If required, the PIS and consent form will be verbally read to the participants by a member of the research team, should they not be able to read English sufficiently to understand the documents. In the unlikely event of the participant being unable to write their own signature, we will ask them to put an X in the appropriate boxes on the consent form. The research team member involved will witness signature the consent form to confirm appropriate consent has been gathered. In this instance, there will also be another witness in addition to the person taking consent.

Reasonable adjustments will also be made for individuals with learning differences - e.g., provide group materials in alternative formats, using pictures as required

#### 8. Storage and analysis of human tissue

N/A for this study.

#### 9. Safety reporting

Any untoward events will be logged on a database, but not reported. This will be for events that are not directly related to the study intervention.

Any adverse events that could be directly related to the intervention, will be logged and reported as per UoB processes

#### 10. Ethical and regulatory considerations

Risk: One of the main ethical considerations for this study, is the potential impact on participants through the GTEP intervention and processing of their traumatic experience. There may be a risk of this intervention temporarily increasing distress or discomfort. To mitigate this risk, there will be breakout rooms available during the sessions for participants to use if they need extra

support from one of the facilitators. All participants will also be offered a catch-up call in between sessions, regardless of whether they have reported distress. As participants will be under the care of the BCPMHS, they will be able to access the duty system should they require further support



outside of the GTEP session times. Participants will be informed of this process during the 1:1 home visit pre-assessment and reminded throughout.

If the participant is identified as needing extra support during the phone calls, then they can be put on the Duty list for a check-in phone call. This might be done by Duty clinician, their care coordinator, any member of staff within the BCPMHS due to have contact with them. This will all be discussed at an MDT and the most appropriate clinician to offer this support will be identified. If the participant continues to report high levels of distress, then they may be offered 1:1 psychology support instead, as per the usual care within the service.

If support is required from the Home Treatment Team, then a referral can be made for this. All decisions regarding extra support will be made as a MDT.

Confidentiality: Given that the group is being completed online, the research team will ensure that participants have access to a confidential space within their homes to engage with the group. This is one of the inclusion criteria for participation in the study. If a participant does not have access to a confidential space, they will be offered 1:1 treatment within the service (depending on their need) rather than the GTEP group. The 1:1 psychology work and corresponding waiting list forms part of the standard care within the BCPMHS.

Ensuring 'treatment as usual': all individuals who participate in the group will still be offered 'treatment-as-usual' within the perinatal service. They will have access to usual support from other disciplines within the multidisciplinary team to ensure that their participation in the group does not get in the way of this. If the participant requires further 1:1 psychological support following the group, then this will be reviewed and discussed during the post-intervention follow-up session. The care team will be informed of the outcome of this decision, and a clinical letter will be sent to their GP.

Access to technology as a barrier: We will ensure that a lack of access to technology (i.e., laptop, internet connection) does not act as a barrier for an individual receiving appropriate support. If an individual does not have access to this, then we will refer them to the digital inclusion project within the Black Country NHS Foundation Trust.

If this is not possible, then the individual will be offered 1:1 support rather than the group, as per standard care in the service.

Informed consent: Before agreeing to take part in the study, potential participants will be provided with a PIS and given the opportunity to discuss the group/research study with members of the team via a phone call. No form of deception will be used in this study and participants will be informed of their right to withdraw at any point. Should they withdraw from the study, they will be offered a 1:1 appointment with a member of the perinatal team to discuss what further psychological support will be needed, and they will be offered 1:1 sessions, if required.

Questionnaire burden: We anticipate that the questionnaires completed at TI and T8 (pre-and-post intervention) will take approximately 20-30 minutes to complete. These can be completed with support from a member of the research team if needed. We anticipate that the PCL-5 outcome measure completed alone at T2, T3, T4, T5, T6 and T7 will take approximately 5-minutes to



complete. Members of the research and clinical team will be available to provide support with completion of questionnaires should the participants require this.

#### 10.1. Assessment and management of risk

Lone working: The 1:1 home visits (session 1 of the intervention) will be completed by a single member of the clinical/research team, in the patient's home. Given this, the team member will follow the lone working policy within the Black Country Perinatal Service.

Risk: There is a risk of the group content (i.e., processing of their traumatic birthing experience) may cause distress and increase risk of participants. If there are any concerns around the safety of a group participant, then a member of the clinical team will contact the participant to discuss this.

Should these concerns remain following this contact, then the process for managing risk within the Black Country Perinatal Service will be followed. This document can be found as part of the Documents Pack for this study.

Any concerns around risk will be documented on the patient's clinical notes. As the GP will have been informed about the participant's engagement with the group, they will also be informed about any concerns regarding a participant's escalating risk via letter.

Safeguarding: All participants will be informed that should a member of the team feel there is a risk of harm to themselves/someone else, then this information will need to be shared with relevant parties. If any safeguarding concerns arise within the group, then the process for managing safeguarding concerns within the Black Country Perinatal Service will be followed. This document can be found as part of the Documents Pack for this study.

Risk to researchers: There is also a potential risk to researchers' wellbeing around exposure to birth trauma experiences. Other members of the research/clinical team will be available for supervision and debrief, if required.

#### 10.2. Research ethics committee (REC) and other regulatory review & reports

Before the start of the project, a favourable opinion will be sought from a REC (NHS REC) for the protocol, informed consent forms and other relevant documents. We will adhere to the following requirements:

- Substantial amendments that require review by NHS REC will not be implemented until that review is in place and other mechanisms are in place to implement this at site
- All correspondence with the REC will be retained
- It is the Cl's responsibility to keep the sponsor updated as required
- The CI will notify the REC and sponsor of the end of the project
- If the project is ended prematurely, the CI will notify the REC and sponsor, including the reasons for the premature termination



Within one year after the end of the project, the CI will submit a final report with the results, including any publications/abstracts, to the REC and sponsor.

10.3.

#### 10.3.1. Regulatory review & compliance

- Before any site can enrol participants into the project, the CI/Principal Investigator or designee will ensure that appropriate approvals from participating organisations are in place.
- For any amendment to the project, the CI or designee, in agreement with the sponsor will submit information to the appropriate body in order for them to issue approval for the amendment. The CI or designee will work with sites (R&D departments at NHS sites as well as the project delivery team) so they can put the necessary arrangements in place to implement the amendment to confirm their support for the project as amended.
- The University of Birmingham's Clinical Research Compliance Team may carry out compliance visits to monitor adherence with applicable standards and regulations.

#### 10.3.2. Amendments

Any amendments to the protocol will be completed by the CI. Decisions about whether an amendment is substantial or non-substantial will be decided by the CI and PI, and other members of the research team stated above. Amendment history will be tracked by having multiple versions of the protocol document, with the file names clearly noting the most recent version (e.g., v1.1., 1.2, 1.,3 etc).

#### 10.4. Peer review

This protocol has been reviewed by staff members within the Black Country Perinatal Mental Health Service and at the University of Birmingham.

It will also be reviewed by the Research and Development Team within the Black Country NHS Foundation Trust.

#### 10.5. Patient & public involvement

The BCPMHS have run a preliminary GTEP group (not involved in the research project) to gather initial feedback on the acceptability of the group for use with a birth trauma population. Based on feedback from participants in this group, the following decisions have been made about the project:

- The number of online sessions increased from 4 to 6 sessions. These six sessions will include three stabilisation sessions and three processing sessions. This will allow more time for stabilisation techniques to be practised and developed. It will also allow time to build relationships between group members and facilitators, and hopefully promote a sense of safety within the group.
- More stringent screening procedures regarding participant suitability. This includes assessing potential participant's presentation in terms of their ability to tolerate a group setting. Participants presenting with high levels of anxiety about the group and/or high levels of dissociation may not be appropriate for the group and will be offered 1:1 support instead.



We have also sought informal feedback from services that have run GTEP groups in other regions, through the GTEP Special Interest Group (SIG).

#### 10.6. Protocol compliance

Accidental protocol deviations can happen at any time. They must be adequately documented on the relevant forms and reported to the CI and Sponsor immediately Significant deviations from the protocol which are found to frequently recur are not acceptable; these will require immediate action and could potentially be classified as a serious breach.

#### 10.7. Data protection and confidentiality

All investigators and site staff must comply with the requirements of the Data Protection Act 2018 with regards to the collection, storage, processing and disclosure of personal information and will uphold the Act's core principles.

#### Data management:

Throughout the project, and afterwards, the data will be stored in line with data protection regulations (i.e. UK GDPR & the Data Protection Act, 2018).

Participant's contact details (including phone number and email address) will be required to arrange the 1:1 home visit (session 1 of the intervention) and send out Zoom links for the GTEP groups sessions. They will also be required to provide a summary of the research findings to the participants, should they request this. This information will be stored on Rio, as per service standards. We will also access demographic information from Rio. There will be a box on the consent form for participants to confirm they are happy for their Rio data to be used for this purpose.

As the worksheets will be completed by participants at their homes during the online sessions, they can either keep them or we can destroy them (e.g., shredding) if they would prefer.

The outcome measures will be completed, and stored on Rio, as per service standards. The numerical participant data (e.g., questionnaire scores) will also be transferred to a password protected database, which will be stored on a secure shared drive within the BCPMHS. Only members of the research team involved with this project will be able to access the database. While we require the data to be identifiable (e.g., to update the data following each session), the participants will be given a participant number on the database and a separate document linking participant number to individual will be created and stored separately to the database. Only team members directly involved in the research study will be able to access this information. Once we no longer require data to be identifiable, a separate spreadsheet without any identifiable information will be created, and any identifiable data will be deleted. For example, we will replace 'date of birth' to 'age by nearest year'. Should data need to be taken 'off site' (e.g., from the BCPMHS shared drive), all identifiable data will be removed. The data will be stored on the BCPMHS shared drive during data collection, and then be securely transferred to the UoB Research Data Store for analysis. Should this database be taken off site (e.g., for data analysis at UoB), all identifiable information will be removed.

The consent forms from MS Forms will be uploaded to Rio as part of their record, so will remain on the clinical record. They will also be kept as part of the research file / data, which will be kept at the University of Birmingham for 10 years.



Data will be kept on the University of Birmingham Research Data Store (RDS) which is backed-up and encrypted. The data will be accessed by the research team only. The research data will be owned by the University of Birmingham.

Data about session attendance will be captured on Rio, as per service standards.

The anonymised databases will be kept for up to 10 years following the end of study/publication. The data stored on the NHS site will be destroyed once the data has been transferred to UoB. The questionnaire data will remain on the participant's Rio records, as per standard practice within the service.

The only individuals able to access the participant's personal data (aside from their usual care team within the perinatal service), will be the research team members.

#### 10.8. Indemnity

The University of Birmingham has in force a Public Liability Policy and/or Clinical Trials Policy which provides cover for claims for 'negligent harm' and the activities here are included within that coverage.

#### 10.9. End of study and archiving

The data will be archived on the University of Birmingham's BEAR archive. Data will be anonymised prior to archiving to ensure there is no patient identifiable information. Data will be kept for up to 10 years following the end of the study/publication.

#### 10.10. Access to the final dataset

The researchers named in this document will have access to the final dataset.

#### 11. Dissemination policy

#### 11.1. Dissemination policy

The data arising from this project will be jointly owned by the Black Country NHS Foundation Trust and the University of Birmingham. On completion of the project, the data will be analysed and tabulated and a final report prepared.

The investigators will have the right to publish the data at the end of the study.

Study participants will notify us via the consent form if they wish to be informed of the results of the study, by provision of the publication. This will be disseminated to them via email, and they will have given consent for their email addresses to be used for this purpose.

#### 11.2. Authorship eligibility guidelines and any intended use of professional writers

The members of the research team outlined in this protocol document will be granted authorship on the final report. Order of authorship will be determined by level of responsibility in this project.



- Ayano, G., Lin, A., Dachew, B. A., Tait, R., Betts, K., & Alati, R. (2022). The impact of parental mental health problems on the educational outcomes of their offspring: Findings from the Raine Study. *Australian & New Zealand Journal of Psychiatry*, *56*(5), 510–524. <a href="https://doi.org/10.1177/00048674211025633">https://doi.org/10.1177/00048674211025633</a>
- Ayers, S., Wright, D. B., & Thornton, A. (2018). Development of a Measure of Postpartum PTSD:

  The City Birth Trauma Scale. *Frontiers in Psychiatry*, 9.

  <a href="https://doi.org/10.3389/fpsyt.2018.00409">https://doi.org/10.3389/fpsyt.2018.00409</a>
- Barkham, M., Bewick, B., Mullin, T., Gilbody, S., Connell, J., Cahill, J., Mellor-Clark, J., Richards, D., Unsworth, G., & Evans, C. (2013). The CORE-10: A short measure of psychological distress for routine use in the psychological therapies. *Counselling and Psychotherapy Research*, 13, 3–13. https://doi.org/10.1080/14733145.2012.729069
- Birth Trauma and Post Natal PTSD PTSD UK. (n.d.). Retrieved 13 March 2024, from <a href="https://www.ptsduk.org/what-is-ptsd/causes-of-ptsd/post-natal-ptsd/">https://www.ptsduk.org/what-is-ptsd/causes-of-ptsd/post-natal-ptsd/</a>
- Blevins, C. A., Weathers, F. W., Davis, M. T., Witte, T. K., & Domino, J. L. (2015). The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. *Journal of Traumatic Stress*, 28(6), 489–498. <a href="https://doi.org/10.1002/jts.22059">https://doi.org/10.1002/jts.22059</a>
- Brockington, I. F., Oates, J., George, S., Turner, D., Vostanis, P., Sullivan, M., Loh, C., & Murdoch, C. (2001). A Screening Questionnaire for mother-infant bonding disorders. *Archives of Women's Mental Health*, *3*(4), 133–140. <a href="https://doi.org/10.1007/s007370170010">https://doi.org/10.1007/s007370170010</a>
- Busse, M., Stromgren, K., Thorngate, L., & Thomas, K. A. (2013). Parent Responses to Stress: PROMIS in the NICU. *Critical Care Nurse*, *33*(4), 52–60. <a href="https://doi.org/10.4037/ccn2013715">https://doi.org/10.4037/ccn2013715</a>
- Chiorino, V., Cattaneo, M. C., Macchi, E. A., Salerno, R., Roveraro, S., Bertolucci, G. G., Mosca, F., Fumagalli, M., Cortinovis, I., Carletto, S., & Fernandez, I. (2020). The EMDR Recent Birth



Trauma Protocol: A pilot randomised clinical trial after traumatic childbirth. *Psychology & Health*, 35(7), 795–810. https://doi.org/10.1080/08870446.2019.1699088

- Dickinson, C., Vangaveti, V., & Browne, A. (2022). Psychological impact of neonatal intensive care unit admissions on parents: A regional perspective. *Australian Journal of Rural Health*, 30(3), 373–384. https://doi.org/10.1111/ajr.12841
- Ertan, D., Hingray, C., Burlacu, E., Sterlé, A., & El-Hage, W. (2021). Post-traumatic stress disorder following childbirth. *BMC Psychiatry*, 21(1), 155. <a href="https://doi.org/10.1186/s12888-021-03158-6">https://doi.org/10.1186/s12888-021-03158-6</a>
- Farrell, D., Moran, J., Miller, P. W., Knibbs, L., Papanikolopoulos, P., McGowan, I., Mattheß, C., & Kiernan, M. D. (2023). Group early intervention eye movement desensitization and reprocessing therapy as a video-conference psychotherapy with frontline/emergency workers in response to the COVID-19 pandemic in the treatment of post-traumatic stress disorder and moral injury—An RCT study. *Frontiers in Psychology*, 14. <a href="https://doi.org/10.3389/fpsyg.2023.1129912">https://doi.org/10.3389/fpsyg.2023.1129912</a>
- Kjerulff, K. H., Attanasio, L. B., Sznajder, K. K., & Brubaker, L. H. (2021). A prospective cohort study of post-traumatic stress disorder and maternal-infant bonding after first childbirth.



Journal of Psychosomatic Research, 144, 110424. https://doi.org/10.1016/j.jpsychores.2021.110424

- Lehnung, M., Shapiro, E., Schreiber, M., & Hofmann, A. (2017). Evaluating the EMDR Group Traumatic Episode Protocol With Refugees: A Field Study. *Journal of EMDR Practice and Research*, 11(3), 129–138. https://doi.org/10.1891/1933-3196.11.3.129
- Manning, C., & Gregoire, A. (2009). Effects of parental mental illness on children. *Psychiatry*, 8(1), 7–9. https://doi.org/10.1016/j.mppsy.2008.10.012
- MBRRACE-UK. Saving Lives, Improving Mothers' Care State of the Nation Surveillance Report: Surveillance findings from the UK Confidential Enquiries into Maternal Deaths 2019-21. Oxford: National Perinatal Epidemiology Unit, University of Oxford 2023
- Pink, J., Ghomi, M., Smart, T., & Richardson, T. (2022). Effects of EMDR Group Traumatic Episode Protocol on Burnout Within IAPT Healthcare Professionals: A Feasibility and Acceptability Study. *Journal of EMDR Practice and Research*, 16(4), 215–227. https://doi.org/10.1891/EMDR-2022-0029
- Roberts, A. K. P. (2018). The effects of the EMDR group traumatic episode protocol with cancer survivors. *Journal of EMDR Practice and Research*, 12(3), 105–117. <a href="https://doi.org/10.1891/1933-3196.12.3.105">https://doi.org/10.1891/1933-3196.12.3.105</a>
- Shapiro, E (2013). "The EMDR Group Traumatic Episode Protocol." Presentation to the EMDR Turkey Conference, Istanbul, Turkey.
- Shapiro, E., & Laub, B. (2008). Early EMDR Intervention (EEI): A Summary, a Theoretical Model, and the Recent Traumatic Episode Protocol (R-TEP). *Journal of EMDR Practice and Research*, 2(2), 79–96. <a href="https://doi.org/10.1891/1933-3196.2.2.79">https://doi.org/10.1891/1933-3196.2.2.79</a>
- Tsouvelas, G., Chondrokouki, M., Nikolaidis, G., & Shapiro, E. (2019). A vicarious trauma preventive approach. The Group Traumatic Episode Protocol EMDR and workplace affect in



professionals who work with child abuse and neglect. 2, 130–138. https://doi.org/10.26386/obrela.v2i3.123

- Weiner, B.J., Lewis, C.C., Stanick, C. *et al.* Psychometric assessment of three newly developed implementation outcome measures. *Implementation Sci* **12**, 108 (2017). https://doi.org/10.1186/s13012-017-0635-3
- Yurtsever, A., Konuk, E., Akyüz, T., Zat, Z., Tükel, F., Çetinkaya, M., Savran, C., & Shapiro, E.
  (2018). An Eye Movement Desensitization and Reprocessing (EMDR) Group Intervention for Syrian Refugees With Post-Traumatic Stress Symptoms: Results of a Randomized Controlled Trial. Frontiers in Psychology, 9. <a href="https://doi.org/10.3389/fpsyg.2018.00493">https://doi.org/10.3389/fpsyg.2018.00493</a>



- 13. Appendices
- 13.1. Appendix 1 - required documentation
- 13.2. Appendix 1a - GTEP Protocol

### **SCRIPT: Group Traumatic Episode Protocol**

this symbol refers to notes only- do not read aloud

#### Script:

'Before starting, you will need colored pencils, felt tips or crayons; a wristband or sticker on your mobile phone, or some other unfamiliar object you wear or carry around which can act as a present focus reminder to check your stress level during the day'.

#### Script:

'You have had a disturbing experience recently which may have affected you in different ways. The work that we will do here today can help your body know that it is safe to feel calmer in this moment and to regain your balance. First we are going to practice the Four Elements exercise'.

'I will also be asking you later to do some Butterfly Hugs or Gorilla Beats/ Chest Taps to strengthen positive connections. Let's try this now'



Demonstrate Butterfly Hugs and Chest Taps/ Gorilla Beats



### Step 1 - Present Safety

#### Script:

'Look at your wristband or sticker and then notice how much stress/anxiety or tension you feel right now on a scale of zero (low) to 10 (high) and write it in the small circle in the yellow Step 1 box next to where it says 'before'.



Show where the Step 1 yellow box is on lower right side of worksheet

#### Script:

'Starting with your feet, we begin with the first element -Earth. Place both feet on the ground, feel the ground and the chair supporting you ....... take a minute to 'land', to take 'time out', to be here, now ......Look around and notice 3 things you did not notice before...... What 3 things do you see? .... ... Now notice what you hear ...... what else?) .... you are here, now .... and you are as safe as can be in this moment.

#### Script:

'Going up your body for the second element,- Air. Notice your breathing ...... now breathe in through your nose letting the air go all the way to your stomach as you count 4 seconds (1...2...3....4) gently hold for 2 seconds (1...2) and then breathe out for 4 seconds (1...2...3...4) Let's take a minute for about 6 deeper slower breaths like this......without any effort, just breathing more deeply and slowly....come back to yourself, to your centre....



#### Script:

'Continue up your body to the third element - Water. Is your mouth dry or do you have saliva? When you are anxious or stressed, your mouth often dries up, but when you are making saliva it is a sign that you are relaxing ...... Take a minute or two to make more and more saliva .... you can imagine the taste of your favourite food, or stimulate the glands at the side of your neck behind your ears. As you do this you may also notice that you have more and more focus and control of your thoughts and body'

#### Script:

'With your feet on the ground, breathing more deeply and slowly; making more and more saliva we move to the fourth element- Light........Bring up an image of a real or imagined place, situation, activity or person that helps you to feel calm and as safe as you can be now. Let's call this your safe or calm place....... In the Step 1 yellow box draw and/or write something that reminds you of this safe or calm place,..., a sketch, symbol or words ....... Notice what you feel when you connect to it and how you feel in your body.' *Give a minute to do this* 

#### Script:

'Keep noticing how you feel in your body when you focus on your safe or calm place....... Give it a name.......and strengthen the connection with a long set of slow Butterfly Hugs as you say the name and focus on your safe place....... Look at your wristband (or sticker) again and notice how much stress you feel now from zero (low stress) to 10 (high stress) and write it in the small circle in the step 1 box next to where it says 'after'.

Who would like to share their safe or calm place?

#### Script:

Practice the Four Elements exercises several times a day. Every time you notice your wristband (or sticker), monitor your stress level from 0-10 and then try to reduce it at least by 1 or 2. After a week or two you may be able to calm yourself more easily just by looking at and touching the object you have chosen. As you practice the Four Elements, your body will find more ways to notice the moments when it is safe to feel calm".



**Note for Group Leader** 

Screen for difficulty in reducing (0 to 10) distress levels. A stress level of 7 or more after the Four Elements exercises indicates a need for further stabilization and preparation before continuing with part two and the remaining steps, or referral.

When continuing the next day or later, begin by briefly reviewing the Four Elements exercise.





# Step 2 – The Start of the Difficult Time

#### Script:

'What we will be doing next can help your natural system digest the things that are still disturbing you from this difficult time. The period of time starting from the date it began to the date today, and even thinking ahead to the future is called the trauma episode.

This exercise will help you to regain your balance. Gradually you can begin feeling as calm, and safe as you can be in this moment.

While you are sitting here safely .... ...with your feet on the ground ....... just notice whatever you notice .....images, thoughts, feelings, body sensations, from the memories of your difficult experiences ......Let's begin by writing the date today here in the Step 1 yellow box, in the circle marked NOW / HERE on the lower right side.



Show where to write the date today in the Step 1 yellow box

#### Script:

'Now write the approximate date of when the difficult time started in the step 2 grey box in the circle marked THERE / THEN on the lower left side.



Show where to write the date in the Step 2 grey box

#### Script:

'Write a headline and/or draw something to represent this initial traumatic event or beginning of the trauma episode. A headline word or words, and/or symbol or sketch.



Pause for group to do this

Rate from 0 to 10 the level of disturbance you feel now, where zero means you can think about it and remain calm and 10 is the highest you know and write it in the small circle in the top left of the step 2 box.'



Show where to write the SUD (0-10). NOTE: No sharing of trauma material




# Step 3 - Good Memory

# Script:

'Remember a time or a moment, when you felt really good about yourself, where you felt whole ......What first comes to mind? ...... Focus only on the good parts of the memory ...... Notice the feelings and body sensations that go with this good memory ......



Show where step 3 green box is on the top left side of the worksheet

# Script:

In the Step 3 green box on the top left side of the worksheet - draw or write something that reminds you of this good memory ....... a sketch, symbol or words......Notice your feelings and body sensations when you connect to the good memory...... Let's strengthen this connection with a long set of slow Butterfly Hugs for 30-40 seconds'......



Demonstrate slow Butterfly Hugs

### Script:

'Keep noticing the feelings and sensations in your body when you focus on your good memory ...... Give it a name and write it down next to the word 'Heading' in the Step 3 box....... Say the name and focus on that good memory and let us strengthen this connection with another long set of slow Butterfly Hugs.

Who would like to share their good memory?



# Step 4 – Positive Thoughts for the Future

### Script:

'Now we move across to the Step 4 pink box on the top right side of the worksheet



Show where Step 4 pink coloured box is on top right side of worksheet

# Script:

'Looking back at this difficult episode, how would you like to think about yourself? Here is a list of suggestions. Mark which of these ways make some sense to you.......Draw or write any other thoughts or pictures of how you would like to see yourself in the future? ......

Who would like to share their positive thought about the future?







# Step 5 – Distancing disturbance (focused processing)

Explanation how to find a Point of Disturbance (PoD) through the Google Scan

## Script:

'We have learned that tapping left to right like this on your worksheet while following with your eyes can help to give distance from a disturbing memory and help you to feel calmer. We still remember it has happened, but it feels further away and sometimes it doesn't feel as disturbing anvmore.'

'Before we start, first I'd like to show you how we find the disturbing parts of the memory we will work on, then we can do it together. I'll be asking you to tap the circle with the date today (in the Step 1 yellow box) and then with the same hand move across the page and tap the circle with the date then (in Step 2 grey box). Continue tapping side to side at a steady pace, making sure you look at your hand as you do this without moving your head.



Demonstrate tapping between the two date boxes

# Script:

'As you tap from side to side at your own pace and look at your hand, think about or scan the whole episode in your mind, from all that has happened from just before it began, up to today and even into the future (like using Google-Search on a computer).

Search for anything still disturbing related to the episode. Memories may come up in no particular order ...... When you find something, stop ...... and draw or write something briefly to represent this disturbing part in the centre of the worksheet in the Step 5 bottom box marked as PoD1 (PoD means Point of Disturbance).'



Show where PoD 1 blue box is located in lower middle section of worksheet

# Script:

Now let's begin the "Google-Search" or scan (date today...date then).....



Wait for all the group to find a PoD and briefly sketched or written in PoD1 ...

'Notice how strong that disturbance feels now from (low) 0 to 10 (high) where zero means you can think about it and remain calm and ten means it's the highest you can imagine. Write this number down in the circle next to PoD1.





# Beginning of PoD processing

<u>Script:</u>
"Touch PoD1 in the step 5 box."



Show where the circle is located on worksheet

### Script:

'Focus on the part that is still disturbing; notice whatever you are thinking, feeling and sensing in your body.

In a moment I will ask you to tap the date today circle at the bottom of the Step1 yellow box and then tap the disturbing part in PoD1 and back again to the date today, like this......Look at your hand going back and forth while you tap... keep tapping as fast as your eyes can comfortably go until I ask you to stop



Demonstrate tapping back and forth between the date today and PoD1

'Let's begin tapping back and forth at your own pace until I ask you to stop....



Time for about 20-30 seconds

### Script:

"Stop. Take a deep breath ...... and let it go. Notice whatever images, thoughts, feelings, or body sensations come up.'

# Script:

'Let's do a second set of tapping as before. Tap date today then Pod 1....



Time for 20-30 seconds

## Script:

'Stop. Take a deep breath ...... and let it go. Notice whatever images, thoughts, feelings, or body sensations come up.'

## Script:

And a third set. Tap date today then Pod 1....



Time for 20-30 seconds

"Stop. Take a deep breath ...... Notice whatever images, thoughts, feelings, or body sensations come up.'

'Re-focus on this upsetting part in PoD1 and check how disturbing it feels for you now, from 0 to 10, where zero means that you can think about it and remain calm and 10 is the highest you know ...... Write this number in the circle at the **top** of the row in PoD1.





# Script:

Continue with a **fourth** set. Tap date today then PoD1... (Time for 20-30 seconds)

"Stop. Take a deep breath ...... and let it go. Notice whatever images, thoughts, feelings, or body sensations come up."

### Script:

And a fifth set. Tap date today then PoD1 (Time for 20-30 seconds)

'Stop. Take a deep breath ...... and let it go. Notice whatever images, thoughts, feelings, or body sensations come up.'

## Script:

'And now a sixth set. Tap date today then PoD1 (Time for 20-30 seconds)

'Stop. Take a deep breath ...... and let it go. Notice whatever images, thoughts, feelings, or body sensations come up.'

## Script:

'Re-focus on this upsetting part in PoD1 and check how disturbing it feels for you now, from 0 to 10, where zero means that you can think about it and remain calm and 10 is the highest you know Write this number in the **middle** circle in PoD1.



Show where the circle is located on worksheet

#### Script:

Continue with a seventh set. Tap date today then PoD1 (Time for 20-30 seconds)

'Stop. Take a deep breath ...... Notice whatever images, thoughts, feelings, or body sensations come up.'

## Script:

And an eighth set. Tap date today then PoD1 (Time for 20-30 seconds).

'Stop. Take a deep breath ...... Notice whatever images, thoughts, feelings, or body sensations come up.'

# Script:

'And now a ninth set. Tap date today then PoD1 (Time for 20-30 seconds).

'Stop. Take a deep breath ...... Notice whatever images, thoughts, feelings, or body sensations come up.'

## Script:

'Re-focus on this upsetting part in PoD1 and check how disturbing it feels for you now, from 0 to 10, where zero means that you can think about it and remain calm and 10 is the highest you know Write this number in the **bottom** circle in PoD1.







# Second Google Scan for PoD2

## Script:

'Let's check for any other disturbing parts of this difficult time. Tap the date today (in the Step 1 yellow box on the lower right side) and then the date then (in the Step 2 grey box on thelower left side), making sure to look at your hand without moving your head."



Demonstrate tapping between the date today and date then boxes

#### Script:

Let's begin....As you do this, scan (or think about) the whole episode in your mind, all that has happened since it began up to today and even in to the future...

Search for anything still disturbing that is related to the episode. Memories may come up in no particular order.........When you find a disturbing part, draw or write something briefly to represent it in the PoD2 box'



Show where the PoD2 box is located on worksheet

#### Script:

'Notice how strong that disturbance feels now from low (0) to 10 (high). Write this number down in the circle directly to the left of PoD2.



Show where the circle is located on worksheet



Processing of PoD2

### Script:

'Now we will process PoD2. Focus on the part in PoD2 that is still disturbing you. Notice whatever you are thinking, feeling and sensing in your body......and tap the date today circle at the bottom of the Step1 box and then the disturbing part in PoD2



Demonstrate tapping back and forth between the date today and PoD2

## Script:

Let's begin tapping until I ask you to stop (Time for 20-30 seconds).

'Stop. Take a deep breath ...... and let it go. Notice whatever images, thoughts, feelings, or body sensations come up.'

'Let's continue with a second set. Tap date today then PoD2......(Time for 20-30 seconds) "Stop. Take a deep breath ...... and let it go. Notice whatever images, thoughts, feelings, or body sensations come up.



### Script:

'And now a third set. Tap date today then PoD 2 ... (Time for 20-30 seconds)

'Stop. Take a deep breath .......and let it go.... Notice whatever images, thoughts, feelings, or body sensations come up.



Show where the circle is located on worksheet

#### Script:

Continue with a fourth set. Tap date today then PoD2... (Time for 20-30 seconds)

'Stop. Take a deep breath ......and notice what comes up.'

#### Script

And a fifth set ..... tap date today then PoD2 (Time for 20-30 seconds)

'Stop. Take a deep breath ......and notice what comes up.'

#### Script

'And now a sixth set ..... tap date today then PoD2 (Time for 20-30 seconds)

'Stop, Take a deep breath ......and notice what comes up

#### Script

'Re-focus on this upsetting part in PoD2 and check how disturbing it feels for you now, from 0 to 10, where zero means that you can think about it and remain calm and 10 is the highest you know Write this number in the **middle** circle in PoD2.



Show where the circle is located on worksheet

### Script

Let's continue with a seventh set ...... tap date today then PoD2 (Time for 20-30 seconds)

'Stop. Take a deep breath ...... and notice what comes up.'

### Script:

And now an eighth set ..... tap date today then PoD2 (Time for 20-30 seconds)

'Stop. Take a deep breath ......and notice what comes up.

### Script:

'And a ninth set... tap date today then PoD2 (Time for 20-30 seconds)

'Stop. Take a deep breath ..... and notice what comes up.

Script:

'Re-focus on this upsetting part in PoD2 and check how disturbing it feels for you now, from 0 to 10, where zero means that you can think about it and remain calm and 10 is the highest you know Write this number in the **bottom** circle in PoD2.







# Third Google Scan for PoD3

### Script:

'Let's check for any other disturbing parts of this difficult time. Tap the date today (in the Step 1 vellow box on the lower right side) and then the date then (in the Step 2 grey box on thelower left side), making sure to look at your hand without moving your head.



Demonstrate tapping between the date today and date then boxes

# Script:

Let's begin....As you do this, scan (or think about) the whole episode in your mind, all that has happened since it began up to today and even in to the future.

Search for anything still disturbing that is related to the episode. Memories may come up in no particular order....... When you find a disturbing part, draw or write something briefly to represent it in the PoD3 box'



Show where the PoD3 box is located on worksheet

# Script:

'Notice how strong that disturbance feels now from low (0) to 10 (high). Write this number down in the circle directly to the left of PoD3.



Show where the circle is located on worksheet



Processing of PoD3

# Script:

'Now we will process PoD3. Focus on the part in PoD3 that is still disturbing you. Notice whatever you are thinking, feeling and sensing in your body...... and tap the date today circle at the bottom of the Step1 box and then the disturbing part in PoD3



Demonstrate tapping back and forth between the date today and PoD3

Let's begin tapping until I ask you to stop (Time for 20-30 seconds).

# Script:

'Stop. Take a deep breath ........ let it go and notice whatever images, thoughts, feelings, or body sensations come up.

'Let's continue with a second set. Tap date today and PoD3 (Time for 20-30 seconds) Stop. Take a deep breath........ and notice whatever images, thoughts, feelings, or body sensations come up.

Protocol version number & date: v1.1,14/03/2025



# Script:

'And now a third set. Tap date today and PoD 3 (Time for 20-30 seconds)

Stop. Take a deep breath....... and notice whatever images, thoughts, feelings, or body sensations come up.

.

# Script:

Re-focus on this upsetting part in PoD3 and check how disturbing it feels for you now, from 0 to 10, where zero means that you can think about it and remain calm and 10 is the highest you know......Write this number in the circle at the **top** of the row in PoD3.



Show where the circle is located on worksheet

### Script

Continue with a fourth set. Tap date today then PoD3... (Time for 20-30 seconds)

'Stop. Take a deep breath ......and notice what comes up.'

#### Script:

And a fifth set ..... tap date today then PoD3 (Time for 20-30 seconds)

'Stop. Take a deep breath ......and notice what comes up.'

### Script:

'And now a sixth set ..... tap date today then PoD3 (Time for 20-30 seconds)

'Stop, Take a deep breath ......and notice what comes up

## Script:

'Re-focus on this upsetting part in PoD3 and check how disturbing it feels for you now, from 0 to 10, where zero means that you can think about it and remain calm and 10 is the highest you know Write this number in the **middle** circle in PoD3.



Show where the circle is located on worksheet

### Script:

Let's continue with a seventh set ...... tap date today then PoD3 (Time for 20-30 seconds)

'Stop. Take a deep breath ...... and notice what comes up.'

### Script:

And now an eighth set ..... tap date today then PoD3 (Time for 20-30 seconds)

'Stop. Take a deep breath ...... and notice what comes up.'

### Script:

'And a ninth set... tap date today to PoD3 (Time for 20-30 seconds)

'Stop. Take a deep breath ...... and notice what comes up.

### Script

'Re-focus on this upsetting part in PoD3 and check how disturbing it feels for you now, from 0 to 10, where zero means that you can think about it and remain calm and 10 is the highest you know Write this number in **bottom** circle in PoD3.







# Step 6-Overall

## Script:

When you think about the whole difficult time/the whole episode, from when it started, up to today, and even into the future ......how disturbing is it for you now from 0 to 10, where zero means you can think about it and remain calm and 10 is the highest you know? Write the number in the small circle in the step 6 purple box on the right side of the worksheet.'



Show where the circle is located in step 6 on the worksheet

'Look at the sentences in the Step 4 pink box (just above step 6) and underline those words that feel most true to you ........ How would you like to think about the whole difficult time/episode now? What have you learned? ..... What are you taking with you from the work that you have done?...... How has this session been for you?'

'Choose the positive words that feel most true to you now........Write this down in the step 6 box ...... Keep repeating them silently to yourself while doing slow Butterfly Hugs or Gorilla Beats to strengthen the connection. Focus on any positive feelings in your body.'

How was that for you? Would anyone like to share? How does your body feel?

# 

# Note for Group Leader

The installation of the positive cognition strengthens the connection between positive thoughts and the disturbing episode. This is not a body scan.



Briefly rehearse the Four Elements and other grounding exercises if needed e.g. Container exercise.

If the Episode SUD level in Step 6 remains high (more than 5) additional G-TEP sessions can be offered or a referral made for individual stabilisation work, G-TEP/R-TEP or Standard Protocol.

# Step 8–Follow-up and screening

Don't forget to follow up. Check Episode SUD level and Positive Cognition.



# **Worksheet to be completed during GTEP Sessions:**





# 13.3. Appendix 2 – amendment history

| The following amendments and/or administrative changes have been made to this protocol since the implementation of the first approved version | | | | |
|---|---|---|---|---|
| Amendment<br>number | Date of amendment | Protocol<br>version number | Type of amendment | Summary of amendment |